CLINICAL TRIAL: NCT05260463
Title: LOQTEQ® Antibacterial Pre-Market Study Randomized, Controlled, Subject-blinded, Multi-center Study of LOQTEQ® Antibacterial Locking Plates in Subjects With Fractures of the Distal Fibula
Brief Title: LOQTEQ® Antibacterial Pre-Market Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: aap Implantate AG (Industry)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: aap001
Record Dates: First submitted 2022-01-11; First posted 2022-03-02 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2024-09

CONDITIONS: Fractures, Open; Fractures, Closed; Surgical Site Infection; Fracture of Fibula
Keywords: Silver-coating; antibacterial; Fibula; Orthopaedic
MeSH Terms: conditions — Fractures, Open; Fractures, Closed; Surgical Wound Infection; Fibula Fractures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Silver-coated Implant (Experimental): The summary description and intended purpose of the investigational device (LOQTEQ® antibacterial silver-coated system) is the same as that of the comparator device (LOQTEQ® 3.5 System (uncoated) system). The investigational device differs from the comparator device in that its surface which has been modified by the addition of an antibacterial coating.
  Interventions: Device: Implantation
- Uncoated Implant (Active Comparator): The summary description and intended purpose of the investigational device (LOQTEQ® antibacterial silver-coated system) is the same as that of the comparator device (LOQTEQ® 3.5 System (uncoated) system) and differes only in the lack of the antibacterial coating.
  Interventions: Device: Implantation

INTERVENTIONS:
Device: Implantation — Fractures of the distal fibula are treated with a trauma implant.

SUMMARY:
aap001 is a randomized, controlled, subject-blinded, multi-center study to show the safety of the LOQTEQ® antibacterial silver-coated system is non-inferior in comparison with the uncoated LOQTEQ® system

DETAILED DESCRIPTION:
Antimicrobial coatings of implants are of interest to reduce infection rate in orthopaedic surgery. Demonstration of clinical effectiveness of such coated implants to obtain market approval is challenging. The objective of this article is to define a design for a randomized controlled trial to evaluate the clinical performance of a silver-coating for locking plates for fracture treatment.

The study design has to respect different criteria, such as feasibility, focus on overall complications, such as functional impairment, fracture healing and infection rates. The study design was defined as randomized, controlled, subject-blinded, multi-center study in subjects with fractures of the distal fibula with a total of 184 patients. A number of 92 patients are planned for each of the two treatment arms with treatment of the fracture with a silver-coated device (first arm) or with an uncoated device (second arm). Inclusion criteria are closed and open fractures of the distal fibula with Gustilo-Anderson type I to Gustilo-Anderson type IIIB type older than 18 years. Primary outcome parameter is the Anticipated Adverse Device Effects (AADE) including all typical complications of this type of injury, such as functional impairment of the affected limb, non-union and infections based on a non-inferiority study design. Also, silver-typical complications, such as argyria, are included. Secondary parameters are infection rates and fracture healing. Follow-up of patients includes five visits with clinical and X-ray evaluations with a follow-up time of 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide voluntary written Informed Consent prior to any study related procedure.
2. Subject aged 18 years and over.
3. Subjects with fractures of the distal fibula.

Exclusion Criteria:

1. Subject unable to give written informed consent, is unlikely to cooperate or is legally incompetent.
2. Subjects with consumptive / malignant primary disease and a life expectancy of less than 12 months.
3. Subjects with a known allergy to silver or any components of the device.
4. Subjects with an already implanted silver-coated device other than the investigational device.
5. History of or ongoing chronic soft-tissue and/or bone and/or implant infection signs at the distal tibia and/or distal fibula (not related to current fracture).
6. Subjects with a possible contraindication for the investigational and comparator devices

   1. infection or inflammation requiring treatment with antibiotics or with positive cultures (not related to current fracture);
   2. acute and chronic osteomyelitis at or close to the surgical field (not related to current fracture);
   3. high anesthesia risk subjects (ASA Physical Status Classification of 4 to 6);
   4. subjects with neurological disorders who cannot follow instructions given by their physician;
   5. subjects with past history of severe medical disorders of extremity which may impact study device efficacy and safety according to investigator's judgment;
   6. severe chronic or acute comorbidity according to investigator's judgement (such as arthritis or neurogenic disorders).
7. Female subjects who are pregnant or lactating at Screening Visit.
8. Females who are of childbearing potential and not taking adequate contraceptive precautions are excluded from the trial. Females of childbearing potential taking acceptable contraceptive precautions according to investigator's judgement can be included.
9. Males with partners who are pregnant or lactating or of childbearing potential and are unwilling to use condoms for the duration of the study. Males who are unable or unwilling to use condoms can be included if partners of childbearing potential taking acceptable contraceptive precautions according to investigator's judgement.
10. Participation in any other study involving an investigational drug or device currently or within the past 3 months.
11. Subject has a significant history of drug/solvent abuse.
12. Subject has a history of alcohol abuse or currently drinks more than 224 g alcohol for men and 112 g alcohol for women per week.
13. Subjects with stage IV vascular disease, i.e. with presence of necrotic tissue at the distal tibia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2025-08-04 (Actual); Study Completion 2025-08-04 (Actual)

PRIMARY OUTCOMES:
Anticipated Adverse Device Effect (AADE) | Implantation until 12 months follow-up
  The primary endpoint for this study is the proportion of subjects with at least one predefined Anticipated Adverse Device Effect (AADE) within 12 months of implantation.

SECONDARY OUTCOMES:
Proportion of subjects with device related infections | Implantation until 12 months follow-up
  Investigate the proportion of subjects with device-related infections occurring after successful implantation of study device and end of the 12-month FU and compare the rate between treatment arms.
Radiographic (X-ray) fracture healing | Implantation until 12 months follow-up
  Investigate fracture healing assessed by local and central reviewer and compare the rate of completely healed subjects between treatment arms.
Hospitalization and nights spent in hospital | Implantation until 12 months follow-up
  Investigate the number of hospitalizations occurring in the first 12 months post-implantation and the nights spent in hospital and compare the numbers between treatment arms.
Change in Ankle-Hindfoot Score (AOFAS) | Implantation until 12 months follow-up
  Investigate the change in AOFAS at each FU visit and compare endpoint between the treatment arms. The change is defined as the difference between AOFAS at the respective FU and the AOFAS at the 1-week FU.
Change in Average Pain at Rest (VAS) | Implantation until 12 months follow-up
  Investigate the change in average pain at rest at each FU visit and compare endpoint between the treatment arms. The Change in Average Pain is defined as the difference between VAS value at the respective FU and the AOFAS at the 1-week FU.
Change in Disability Rating Index (DRI) | Implantation until 12 months follow-up
  Investigate the change in the disability rating index at each FU visit and compare endpoint between the treatment arms. The change in DRI is defined as the difference between DRI at the respective FU and at the 1-week FU.
EQ-5D-5L | Implantation until 12 months follow-up
  Investigate all items assessed in the EQ-5D-5L questionnaire. The changes from Screening will be compared between treatment arms for all FU visits.
Weight bearing | Implantation until 12 months follow-up
  Investigate the proportion of subjects with full weight bearing at each FU visit and compare this endpoint between the treatment arms.
Change in Silver Serum Levels | Implantation until 12 months follow-up
  Investigate the change in silver serum levels at each scheduled FU visit and compare endpoint between the treatment arms. The change in silver serum level is defined as the difference between the respective silver level at the respective FU and the silver level at Screening/Enrollment Visit.
Proportion of subjects with Treatment emergent adverse events (TEAE) | Implantation until 12 months follow-up
  Investigate the proportion of subjects with TEAEs during the 12-month FU and compare the rate between treatment arms.

CONTACTS AND LOCATIONS:
Overall Officials: Volker Alt, Prof. Dr., Study Director — Universitätsklinikum Regensburg
Locations (13):
- Germany (13):
  - Universitätsklinikum Regensburg, Regensburg, Bavaria
  - Unfallkrankenhaus Berlin, Berlin
  - Helios Klinikum Berlin-Buch GmbH, Berlin
  - Städtisches Klinikum Dresden, Dresden
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsklinikum Gießen-Marburg, Giessen
  - Universitätsklinikum Homburg-Saar, Homburg
  - Universitätsklinikum Leipzig, Leipzig
  - Universitätsklinikum Münster, Münster
  - Universitätsklinikum Rostock, Rostock
  - Agaplesion Bethesda Krankenhaus Wuppertal, Wuppertal
  - Helios Universitätsklinikum Wuppertal, Wuppertal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schoder S, Lafuente M, Alt V. Silver-coated versus uncoated locking plates in subjects with fractures of the distal tibia: a randomized, subject and observer-blinded, multi-center non-inferiority study. Trials. 2022 Dec 1;23(1):968. doi: 10.1186/s13063-022-06919-0. PMID 36456987